CLINICAL TRIAL: NCT01512498
Title: Vulvovaginal Graft Versus Host Disease in Women Who Underwent Transplantation Before and After Menarche
Brief Title: Vulvovaginal Graft Versus Host Disease (VV-GVHD) in Women Who Underwent Transplantation Before and After Menarche
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, Senior physician, the clinic for vulvovaginal disorders, Hadassah Mt Scopus, Hadassah Medical Organization
Other Study IDs: MYS-09-HMO-CTIL
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Graft-vs-Host Disease
Keywords: VV GVHD; girls; adolescents; HSCT
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who underwent allogeneic HSCT: Patients who underwent allogeneic HSCT before the age of 18, who are 18 years or older at the time of the study and who are alive.

SUMMARY:
The study will evaluate the prevalence and characteristics of vulvovaginal graft versus host disease (VV- GVHD) in patients who underwent hematopoietic stem cell transplantation (HSCT) as girls or adolescents and will compare the prevalence, characteristics and severity of VV-GVHD before and after menarche.

DETAILED DESCRIPTION:
The phenomenon of vulvovaginal graft versus host disease (VV-GVHD) following hematopoietic stem cell transplantation (HSCT) was first described in 1982 [Corson]. It is characterized by vulvovaginal inflammation, scarring, adhesions and might end with complete vaginal obliteration. Hematopoietic stem cells source for the allogeneic transplantation was found to affect the incidence of VV-GVHD: peripheral blood progenitor cells were associated with an incidence of 50% [Zantomio], while bone-marrow harvested cells were associated with an incidence of 25% [Spinelli].

Due to the high incidence of genital GVHD and its severe consequences we established a clinic designated for post- transplantation patients at the Hadassah University Hospital in Jerusalem. In a two years follow-up we found an incidence of 54% vulvovaginal GVHD in adult patients who attended the clinic, similar to the incidence described in the literature.

The data on VV-GVHD in the literature refers mainly to adult women. As gynecological examination and follow-up is not done routinely in girls and adolescents who are not sexually active, the incidence and characteristics of VV-GVHD in girls and adolescents who underwent HSCT is unknown.

Methods:

Patients who underwent allogeneic HSCT before the age of 18, who are 18 years or older at the time of the study and who are alive will be invited to participate in the study. Those who will be willing to participate will complete questionnaires and undergo physical and gynecological examination. At a single appointment, data will be acquired regarding: age, time from transplantation, current medical status, medications,hormonal status,marital status, sexual function and fertility (pregnancies and deliveries), assessment of sexual development by a pediatric endocrinologist regarding Tunner stages,data regarding possible vulvovaginal involvement, presence and scoring of GVHD in other organs and assessment of patients' well being using the FACT-BMT score.

In order to assess engraftment and degree of chimerism, donor and host-specific DNA markers, using male and female amelogenine gene PCR bands and by STR-PCR assay will be done.

Gynecological exam: in case the patient is sexually active, a complete vulvovaginal exam using a speculum, bimanual exam and transvaginal ultrasound will be done. In case the patient never had sexual intercourse, only external (vulvar) exam and abdominal ultrasound exam will be done.

On exam, the following aspects will be evaluated: vulvar anatomy, vaginal examination for adhesions, fibrosis or stenosis. Vaginal exam will include vaginal pH measurement, saline and 10% potassium hydroxide microscopy, evaluation for the presence of condylomas, Pap smear and vaginal and cervical swab for HPV.

VV-GVHD will be defined according to clinical criteria, which include vulvovaginal anatomic changes, mucosal erosion and inflammation.

Blood samples will be examined for:

hormonal status, measurements of blood Th1/Th2 cytokines and immunoglobulins levels.

Immune reconstitution will be evaluated by quantitative immune reconstitution done using peripheral blood cells. The cells will be analyzed by flow cytometry using fluorescein isothiocyanate antibodies for the absolute counts of various T cells sub populations, B cells, NK and NKT cells.

Additional data regarding age at transplantation, menarchal status at transplantation, sexual activity status at time of transplantation, diagnosis, donor relation, source of cells, number of cells infused, protocol, conditioning regimen, immunosuppressive prophylaxis and occurrence of GVHD in other organs will be acquired by anamnesis and from the patients' files.

ELIGIBILITY:
Inclusion criteria:

* Patients who underwent allogeneic HSCT before the age of 18, who are 18 years or older at the time of the study and who are willing to participate in the study .

Exclusion Criteria:

* not able to comply with the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent allogeneic HSCT before the age of 18, who are 18 years or older at the time of the study and who are alive .
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
incidence of VV- GVHD in patients who underwent HSCT as girls or adolescents. | 1 day
  Patients who underwent HSCT before the age of 18, who are 18 years or older at the time of the study, will be invited for a single appointment evaluation. Time from HSCT will range according to the date of transplantation, varying between 1-30 years.

SECONDARY OUTCOMES:
Prevalence, characteristics and severity of VV-GVHD before and after menarche | 1 day
Effect of sexual intercourse and/or virginity on the clinical manifestations of VV-GVHD in girls and adolescents. | 1 day
Sexual development and maturity in regard to genital anatomy and the presence of VV-GVHD. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Hadassah University Hospital, Jerusalem, ISRAEL
Locations (2):
- Israel (2):
  - Pediatric Hematology Oncology Department, Rambam Hospital, Haifa
  - Hadassah University Hospital, Jerusalem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zantomio D, Grigg AP, MacGregor L, Panek-Hudson Y, Szer J, Ayton R. Female genital tract graft-versus-host disease: incidence, risk factors and recommendations for management. Bone Marrow Transplant. 2006 Oct;38(8):567-72. doi: 10.1038/sj.bmt.1705487. Epub 2006 Sep 4. PMID 16953208
- [Background] Spinelli S, Chiodi S, Costantini S, Van Lint MT, Raiola AM, Ravera GB, Bacigalupo A. Female genital tract graft-versus-host disease following allogeneic bone marrow transplantation. Haematologica. 2003 Oct;88(10):1163-8. PMID 14555313
- [Background] Corson SL, Sullivan K, Batzer F, August C, Storb R, Thomas ED. Gynecologic manifestations of chronic graft-versus-host disease. Obstet Gynecol. 1982 Oct;60(4):488-92. PMID 6750475